CLINICAL TRIAL: NCT07352709
Title: Understanding the Effect of Feedback on Ventilation Performance of Rescuers in a Simulation Trial
Brief Title: Ventilation Performance and Feedback Simulation Trial
Acronym: VENT-SIM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Betty Yang, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STU20252216
Record Dates: First submitted 2025-12-17; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Out-of-hospital Cardiac Arrest (OHCA)
Keywords: ventilation during resuscitation; CPR; emergency medical services
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Intervention Model Description: Randomized crossover trial with an embedded 2x2 factorial design. We will compare real-time visual feedback (with vs without) primarily and CPR strategy (interrupted compressions and ventilations given during pauses vs continuous compressions and ventilations given interposed). Each provider will serve as their own control and crossover midway on feedback. Each provider will provide ventilations for 5 minutes per arm, for a total of 20 minutes. Each provider will be randomized to the sequence of feedback and CPR strategy, using randomized block design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard CPR with interrupted compressions with feedback (Experimental)
  Interventions: Other: Real-time feedback
- Standard CPR with interrupted compressions without feedback (No Intervention)
- Continuous chest compressions with feedback (Experimental)
  Interventions: Other: Real-time feedback
- Continuous chest compressions without feedback (No Intervention)

INTERVENTIONS:
Other: Real-time feedback — Visual feedback provided on volumes insufflated and expired
  Arms: Continuous chest compressions with feedback; Standard CPR with interrupted compressions with feedback

SUMMARY:
The study "Understanding the Effect of Feedback on Ventilation Performance of Rescuers in a Simulation Trial" will address treatments administered by Emergency Medical Services (EMS) during cardiopulmonary resuscitation (CPR) in simulated out-of-hospital cardiac arrest (OHCA). The investigators propose a randomized controlled trial among EMS responders to compare quality of rescue breathing performance with and without real-time feedback, along with evaluating CPR strategies (providing rescue breathing during pauses interrupting chest compression vs rescue breathing during uninterrupted chest compressions). The goal of this trial is to learn if visual feedback improves the ability of rescuers to deliver a specified amount of air. The main questions the study aims to answer are:

* Does real-time visual feedback improve ventilation performance and the ability of rescuers to provide a specified amount of air?
* Will different CPR strategies change the effect of feedback on performance? Researchers will compare real-time feedback to no feedback (not showing the visual feedback) to see if real-time feedback works to improve performance.

Rescuers will:

* Deliver assisted ventilation breaths to a mannequin with and without feedback with two different CPR strategies in one session.
* Fill out a survey about the experience level.

DETAILED DESCRIPTION:
The study "Understanding the Effect of Feedback on Ventilation Performance of Rescuers in a Simulation Trial" will address treatments administered by Emergency Medical Services (EMS) during cardiopulmonary resuscitation (CPR) in simulated out-of-hospital cardiac arrest (OHCA). Guidelines have recommended delivering assisted rescue breaths at a volume of 500-600 mL or until chest rise. Current standard of practice for CPR strategies is either to deliver 2 rescue breaths during a pause after 30 chest compressions or 1 rescue breath at a rate of 10 breaths per minute during continuous chest compressions. Scientific studies have shown that EMS clinicians have administered rescue breath volumes and rates that can be too high or too low; both extremes can be harmful to patient lungs and outcomes. Despite guideline recommendations on volumes, EMS performance and adherence to specific targets with real-time feedback have not been well tested and compared between the two CPR strategies. Thus, the goal of this trial is to learn if visual feedback improves ventilation performance of rescuers, and assess whether this differs when comparing the two CPR strategies.

The study will address two primary aims:

Aim 1. Test whether adherence to specific targets improves with real-time visual feedback during CPR. The hypothesis is that real-time visual feedback will result in a higher rate of adherence to specific targets.

Aim 2. To compare adherence to specific targets during CPR strategy of 30:2 chest compressions: rescue breaths versus continuous chest compressions and rescue breaths. The hypothesis is that rescue breaths delivered during interrupted chest compressions will result in better compliance with specific targets than those delivered during continuous chest compressions.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Credentialed EMS

Exclusion Criteria:

* EMS Instructor
* Inactive EMS role

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2031-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of guideline compliant ventilations | 20 minutes
  proportion of ventilations within the target ventilation parameters (tidal volume 500-600 mL)

SECONDARY OUTCOMES:
Volume insufflated | 20 minutes
Volume expired | 20 minutes
Ventilation rate | 20 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided